CLINICAL TRIAL: NCT02566915
Title: Effects of Expiratory Positive Airway Pressure on Dyspnea and Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Exhalation Valve on the Lack of Air and Exercise Tolerance in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-0067
Record Dates: First submitted 2015-09-25; First posted 2015-10-02 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPET submaximal without EPAP (No Intervention): Will be collected clinical and anthropometric data of the participants and they are packaged in self-evaluation form. Evaluation of pulmonary function at rest will be rescued from patient charts. When carried out for over six months, will be repeated by the researchers. Patients will conduct incremental CPET of 5-10W/min limited by symptoms (FEV1 <1L-5W or FEV1> 1L-10W) (Visit 1). After a period of 2-7 days the CPET will be performed submaximal with 75% of the peak load reached in the incremental CPET (visits 2-3). During the visit without EPAP will be maintained using the facial mask applied without resistance.
- CPET submaximal with EPAP (Experimental): Will be collected clinical and anthropometric data of the participants and they are packaged in self-evaluation form. Evaluation of pulmonary function at rest will be rescued from patient charts. When carried out for over six months, will be repeated by the researchers. Patients will conduct incremental CPET of 5-10W/min limited by symptoms (FEV1 <1L-5W or FEV1> 1L-10W) (Visit 1). After a period of 2-7 days the CPET will be performed submaximal with 75% of the peak load reached in the incremental CPET (visits 2-3). The application of EPAP (10cmH2O) via face mask (Vital RHDSON Signs®, New Jersey, USA) will be randomized with the help of opaque envelopes to be given in one visit. IC serial measurements will be carried out before, during and immediately after the exercise.
  Interventions: Device: CPET submaximal with EPAP

INTERVENTIONS:
Device: CPET submaximal with EPAP — The expiratory positive pressure is applied through silicone mask (RHDSON Vital Signs®, New Jersey, USA) containing one-way valve and a resistance mechanism expiratory positive expiratory pressure generator adjustable 5-20 cm H2O (Spring Loaded) (Vital Signs® , New Jersey, USA). The mask one headgear will be comfortably adjusted to face being used to prevent air leakage, and the pressure level gradually adjusted to the level of 10 cm H2O.
  Arms: CPET submaximal with EPAP

SUMMARY:
The purpose of this study is to evaluate the effects of the application of Expiratory Positive Airway Pressure (EPAP) on Dynamic Hyperinflation, dyspnea and exercise tolerance in patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Initially will be collected clinical and anthropometric data of the participants, and they are packaged in self-evaluation form. The evaluation of pulmonary function at rest (spirometry, body plethysmography and lung diffusion capacity for carbon monoxide) will be rescued from patient charts. When carried out for over six months, will be repeated by the researchers. Patients will conduct incremental CPET of 5-10W / min limited by symptoms (FEV1 <1L - 5W or FEV1> 1L - 10W) (Visit 1). After a period of 2-7 days the CPET will be performed submaximal with 75% of the peak load reached in the incremental CPET (visits 2 and 3). The application of EPAP (10cmH2O) via face mask (Vital RHDSON Signs®, New Jersey, USA) will be randomized with the help of opaque envelopes to be given in one visit. During the visit without EPAP will be maintained using the facial mask applied without resistance. IC serial measurements will be carried out before, during and immediately after the exercise. Participants will be instructed to maintain the use of long-acting bronchodilator as prescribed by the medical assistant usually before the methodological stages of the study.

ELIGIBILITY:
Inclusion Criteria:

* clinically stable patients without exacerbation of signs in the eight weeks preceding the study
* making use of drug therapy (long-acting bronchodilators)
* able to perform the exercise on the bike
* without other comorbidities that compromise the results exercise
* sign the Informed Consent

Exclusion Criteria:

* associated heart diseases
* diagnosis of asthma
* Oxygen therapy use
* SpO2 <85% at rest
* use of oral corticosteroids or antihistamines
* use of artificial airway
* musculoskeletal dysfunction

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Increased Inspiratory Capacity (IC) through dynamic changes in lung volumes | 1 year
  This technique assumes that the TLC remains unchanged during exercise, even in patients with COPD: thus, changes in IC will reflect in proportional changes in end-expiratory lung volume (EELV). The validity, reproducibility and sensitivity to these interventions have been demonstrated by this technique in patients with COPD, showing a variety of functional abnormalities.
  Before the test, the patients will be familiar with this technique by performing IC maneuvers. They will be instructed to breathe normally during exercise and then, through verbal commands, will conduct a deep breath followed by a relaxed expiration. During inspiration, patients will be encouraged to make every effort.
  IC maneuvers are performed during the rest period are obtained until at least two reproducible efforts, namely within 10% of the highest acceptable value. After that, measurements of IC will be held every two minutes until exhaustion.

SECONDARY OUTCOMES:
Increased exercise tolerance submaximal CPET | 1 year
  To assess exercise tolerance we will compare the final time the two submaximal CPET (with EPAP and without EPAP). In each test, the patient will be encouraged to achieve maximum tolerance and will be instructed to stop the test in the exhaust.
Decreased dyspnea submaximal CPET | 1 year
  To evaluate the sensation of dyspnea the year we will be using the modified Borg scale. This measurement will be held every two minutes during the two submaximal CPET (with EPAP and without EPAP).

CONTACTS AND LOCATIONS:
Overall Officials: Danilo C Berton, Principal Investigator — HCPA/UFRGS; Marli M Knorst, Study Chair — HCPA/UFRGS; Mariane B Monteiro, Study Chair — IPA; Paulo José Z Teixeira, Study Chair — Federal University of Health Science of Porto Alegre; Dulciane N Paiva, Study Chair — University of Santa Cruz do Sul; Dannuey M Cardoso, Study Chair — University of Santa Cruz do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] O'Donnell DE, Gebke KB. Activity restriction in mild COPD: a challenging clinical problem. Int J Chron Obstruct Pulmon Dis. 2014 Jun 4;9:577-88. doi: 10.2147/COPD.S62766. eCollection 2014. PMID 24940054
- [Background] Gagnon P, Guenette JA, Langer D, Laviolette L, Mainguy V, Maltais F, Ribeiro F, Saey D. Pathogenesis of hyperinflation in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Feb 15;9:187-201. doi: 10.2147/COPD.S38934. eCollection 2014. PMID 24600216
- [Background] Silveira L, Teixeira PJ, da Costa CC, de Souza RM, Merola PK, Colombo C, Marques RD, Berton DC. The relationship between fat-free mass index and pulmonary hyperinflation in COPD patients. Respirology. 2014 Nov;19(8):1204-8. doi: 10.1111/resp.12406. PMID 25302758
- [Background] Pessoa IM, Costa D, Velloso M, Mancuzo E, Reis MA, Parreira VF. Effects of noninvasive ventilation on dynamic hiperinflation of patients with COPD during activities of daily living with upper limbs. Rev Bras Fisioter. 2012 Jan-Feb;16(1):61-7. English, Portuguese. PMID 22441230
- [Background] Andersen JB, Qvist J, Kann T. Recruiting collapsed lung through collateral channels with positive end-expiratory pressure. Scand J Respir Dis. 1979 Oct;60(5):260-6. PMID 392747
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Belman MJ, Botnick WC, Shin JW. Inhaled bronchodilators reduce dynamic hyperinflation during exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1996 Mar;153(3):967-75. doi: 10.1164/ajrccm.153.3.8630581.
- [Background] Yan S, Kaminski D, Sliwinski P. Reliability of inspiratory capacity for estimating end-expiratory lung volume changes during exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Jul;156(1):55-9. doi: 10.1164/ajrccm.156.1.9608113. PMID 9230726
- [Background] O'Donnell DE, Lam M, Webb KA. Measurement of symptoms, lung hyperinflation, and endurance during exercise in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1557-65. doi: 10.1164/ajrccm.158.5.9804004. PMID 9817708
- [Background] Mahler DA, Weinberg DH, Wells CK, Feinstein AR. The measurement of dyspnea. Contents, interobserver agreement, and physiologic correlates of two new clinical indexes. Chest. 1984 Jun;85(6):751-8. doi: 10.1378/chest.85.6.751. PMID 6723384
- [Result] Monteiro MB, Berton DC, Moreira MA, Menna-Barreto SS, Teixeira PJ. Effects of expiratory positive airway pressure on dynamic hyperinflation during exercise in patients with COPD. Respir Care. 2012 Sep;57(9):1405-12. doi: 10.4187/respcare.01481. Epub 2012 Feb 17. PMID 22348429
- [Result] Neder JA, Andreoni S, Peres C, Nery LE. Reference values for lung function tests. III. Carbon monoxide diffusing capacity (transfer factor). Braz J Med Biol Res. 1999 Jun;32(6):729-37. doi: 10.1590/s0100-879x1999000600008. PMID 10412551
- [Result] O'Donnell DE, Sanii R, Giesbrecht G, Younes M. Effect of continuous positive airway pressure on respiratory sensation in patients with chronic obstructive pulmonary disease during submaximal exercise. Am Rev Respir Dis. 1988 Nov;138(5):1185-91. doi: 10.1164/ajrccm/138.5.1185. PMID 3059891
- [Result] Nicolini A, Merliak F, Barlascini C. Use of positive expiratory pressure during six minute walk test: results in patients with moderate to severe chronic obstructive pulmonary disease. Multidiscip Respir Med. 2013 Mar 14;8(1):19. doi: 10.1186/2049-6958-8-19. PMID 23497658
- [Result] Soares SM, Oliveira RA, Franca SA, Rezende SM, Dragosavac D, Kacmarek RM, Carvalho CR. Continuous positive airway pressure increases inspiratory capacity of COPD patients. Respirology. 2008 May;13(3):387-93. doi: 10.1111/j.1440-1843.2008.01263.x. PMID 18399861
- See also: Reference values for lung function testes. I.Static volumes. — http://www.scielo.br/pdf/bjmbr/v32n6/3179c.pdf
- See also: Analysis of chest radiography of individuals with COPD and its correlation with functional testing — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0103-51502012000300018
- See also: Dynamic hyperinflation during treadmill exercise testing in patients with moderate to severe COPD — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1806-37132012000100004
- See also: Determining anaerobic threshold through heart rate variability in patients with COPD during cycloergometer exercise — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0103-51502012000400004
- See also: Comparison of the physiological variables in the six-minute walk test and stair-climbing test in patients with chronic obstructive pulmonary disease — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1517-86922012000500002&lng=en&nrm=iso&tlng=en
- See also: Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease — http://www.scielo.br/pdf/jbpneu/v34n12/v34n12a05.pdf